CLINICAL TRIAL: NCT06221384
Title: Comparison of Modified Two-Dimensional and M-mode TAPSE With Transesophageal Echocardiography and M-mode TAPSE With Transthoracic Echocardiography in Pediatric Cardiac Transcatheter Interventions
Brief Title: Transesophageal Echocardiography Transthoracic Echocardiography TAPSE
Acronym: TAPSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, ferdi gülaştı, assistant prof.dr., Aydin Adnan Menderes University
Other Study IDs: 2024-1
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-01

CONDITIONS: We Aim to Compare Modified Tricuspid Annular Plane Systolic Excursion With Tricuspid Annular Plane Systolic Excursion
Keywords: TAPSE; Modified TAPSE; Pediatric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Modified TAPSE (m-TAPSE) is a new method in which TAPSE is measured by taking the difference between the apical and lateral tricuspid annulus distance during diastole and systole. It can be measured using transesophageal echocardiography (TEE) in the mid-esophageal four-chamber (ME 4CH) view and is an alternative easily measurable parameter for intraoperative assessment of RV systolic function as long as optimal imaging quality is achieved.

In this prospective observational study, between 01.02.2024 and 01.01.2025, patients between the ages of 1-18 will undergo transcatheterization procedures using TTE and TEE under anesthesia by a pediatric cardiologist. TAPSE of these patients will be measured by TTE and TEE. TAPSE of the patients will be evaluated with TTE and TOE.

DETAILED DESCRIPTION:
Modified TAPSE (m-TAPSE) is a new method in which TAPSE is measured by taking the difference between the apical and lateral tricuspid annulus distance during diastole and systole. It can be measured using transesophageal echocardiography (TEE) in the mid-esophageal four-chamber (ME 4CH) view and is an alternative easily measurable parameter for intraoperative assessment of RV systolic function as long as optimal imaging quality is achieved.

Our study will begin between 01.02.2024 and 01.01.2025 at Adnan Menderes University Practice and Research Hospital, after receiving the approval of the Ethics Committee of the patients. In this prospective observational study, it was planned to include all patients between the ages of 1 and 18 who underwent transcatheterization procedures using TTE and TEE under anesthesia by pediatric cardiologist. Written and verbal consent will be obtained from the parents/guardians of the patients. Patients will be anesthetized for transcatheter procedures and TAPSE and FAC values will be recorded during TTE and TEE echocardiography for the procedure. Two practitioners will make the measurements and each of their own values will be recorded. After the data collection process for the study is completed; The data will be compared statistically. TTE and TEE values of the patients will be compared among themselves.

All patients will undergo TEE and TTE under general anesthesia with an Echocardiography Device. The values of all parameters will be recorded by taking the average values of three cardiac cycle measurements. Measurement methods will be performed in accordance with the American Society of Echocardiography Guidelines. M-Mode, 2D images, color, pulse, Continuous Wave Doppler and Tissue Doppler measurements will be taken from all subjects complying with standard echocardiographic application methods. TAPSE will be calculated by placing an M-mode cursor across the Tricuspid Annulus and measuring the amount of longitudinal movement at peak systole.

m-TAPSE by TOE: m-TAPSE will be calculated as the 'difference between the apical to lateral tricuspid annular distance' during diastole and systole measured in the ME 4CH view. Within this cycle, the maximum and minimum dimensions will be obtained and the difference will be used to measure m-TAPSE. Longitudinal movement during systole will be measured by performing enhanced Doppler alignment with a modified transgastric RV inlet view and lower tricuspid annular motion.

End-diastolic area (EDA) and end-systolic area (ESA) are the FAC measurements that will be used in the TTE apical four-chamber view, while the same measurement will be made in the TEE four-chamber view, which also shows EDA and ESA.

ELIGIBILITY:
Inclusion Criteria:

* 1- Hastanın 1-18 yaş arasında olması 2- Pediyatrik kardiyak transkataterizasyon işlemi yapılması 3- ASA 1-3 hastalar

Exclusion Criteria:

* 1- Veli veya vasinin onay vermemesi 2- ASA 4 ve üzeri hastalar

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Transcatheterization procedures using TTE and TEE under anesthesia will be performed by pediatric cardiologist between the ages of 1-18.
Sampling Method: Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
echo | 30 minute
  Intraoperatively, TAPSE and modified TAPSE values of patients will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Ferdi Gülaştı, Aydin, Turkey (Türkiye)